CLINICAL TRIAL: NCT00218699
Title: Changing Sexual Behavior in Gay Male Repeat HIV Testers: A Randomized Trial of a Single Session Counseling Intervention
Brief Title: Pre-HIV Test Counseling Intervention to Reduce HIV Infection Risk Behavior in Men Who Are Not HIV Infected
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: James W. Dilley, MD/Principal Investigator, University of California, San Francisco - Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH065138 (NIH); R01MH065138 (NIH); DAHBR AZ-Q
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections
Keywords: HIV; MSM Men Who Have Sex with Men; Men Who Have Sex With Men; Cognitive-Behavioral; HIV Counseling and Testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention

SUMMARY:
This study will evaluate the effectiveness of a single specialized pre-test counseling session in reducing HIV infection risk behavior in men who are not HIV infected.

DETAILED DESCRIPTION:
In San Francisco, HIV infection rates among men who have tested for HIV three or more times is almost triple the HIV infection rates of all other testers. Past research has shown that HIV uninfected gay and bisexual men who receive counseling are less likely to engage in high-risk sexual behavior. Counseling provided by trained mental health professionals within a clinical study setting helped individuals identify and re-evaluate their "self-justifications," which are their thoughts, attitudes, and beliefs when deciding to engage in unprotected sex. This study will focus on implementing a "real-world" counseling intervention designed specifically for men who are at the greatest risk of becoming infected with HIV: men who engage in high-risk sexual activity with other men and who repeatedly test for HIV. This specialized intervention will be administered by trained paraprofessional counselors during a pre-test counseling session prior to an HIV test. The purpose of this study is to evaluate the effectiveness of the specialized pre-test counseling intervention versus a standard pre-test counseling intervention in promoting safer sexual activity among HIV uninfected men. The men will have reported having unprotected sex with males of unknown HIV status or known HIV infection.

This 12-month study will enroll 300 men who will be recruited upon scheduling an anonymous HIV test at the participating clinic. Participants will be randomly assigned to receive either the enhanced pre-test counseling session or a standard pre-test counseling session prior to an HIV test. Outcome measurements will be assessed 6 and 12 months after the counseling session and will include self-reports of unprotected anal sex with non-primary partners and reported satisfaction levels with the pre-test counseling.

ELIGIBILITY:
Inclusion Criteria:

* History of two or more HIV antibody tests prior to study entry
* History of at least one episode of unprotected anal intercourse (receptive or insertive) within 12 months prior to study entry

Exclusion Criteria:

* History of injection drug use within 12 months of study enrollment
* Insufficient proficiency in English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2002-08; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV infection risk behavior; measured at Months 6 and 12 | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James W. Dilley, MD, Principal Investigator — UCSF AIDS Health Project; William J. Woods, PhD, Principal Investigator — UCSF Center for AIDS Prevention Studies
Locations (1):
- UCSF AIDS Health Project, San Francisco, California, United States